CLINICAL TRIAL: NCT05251987
Title: Comparison of High PD1+ T Cell and Low PD1+ T Cell Expression in Peripheral Blood for Cardiac Function Prognosis in Patients With Acute Myocardial Infarction
Brief Title: Comparison of PD1+T Cell Expression in Peripheral Blood for Cardiac Function Prognosis in Patients With Acute MI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0725
Record Dates: First submitted 2022-01-17; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-10

CONDITIONS: PD1; Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High PD1+ T Cell Expression: high PD1+ T cell expression in peripheral blood
  Interventions: Biological: PD1+ T Cell Expression
- Low PD1+ T Cell Expression: low PD1+ T cell expression in peripheral blood
  Interventions: Biological: PD1+ T Cell Expression

INTERVENTIONS:
Biological: PD1+ T Cell Expression — The expression of PD1+ T cells was detected by flow cytometry in peripheral blood

SUMMARY:
Comparison of high PD1+ T cell and low PD1+ T cell expression in peripheral blood for cardiac function prognosis in Patients with acute myocardial infarction

DETAILED DESCRIPTION:
Myocardial infarction is a serious common disease in human beings. Although many patients with acute myocardial infarction survive with the improvement of medical technology in recent years, studies have shown that cardiac remodeling caused by myocardial remodeling after myocardial infarction can still lead to heart failure. Severe heart failure is the main cause of death. Myocardial infarction is a process in which multiple cells interact and participate in post-infarction repair. The pathophysiological processes include early angiogenesis, myocardial compensatory hypertrophy and chronic rational myocardial remodeling and fibrosis. Accordingly, how immune inflammatory cells regulate angiogenesis and fibroblast activation during chronic myocardial remodeling are important therapeutic targets for improving the prognosis of myocardial infarction.Each phase after myocardial infarction has its characteristic pathophysiological changes. Studies have shown that immune inflammatory cells T cells are involved in the whole process of regulating the repair of myocardial infarction. Immune studies have shown that PD1/PD-L1, as a second stimulation signaling pathway besides the antigen TCR of T cells, has the ability to inhibit THE activity of T cells, so the inhibition of PD1/PD-L1 has become a research hotspot in the field of tumor therapy. A large number of studies have focused on the regulation mechanism of PD1/PD-L1 signaling pathway in tumor immune cell activity. Regarding PD1/PD-L1 as the mechanism of immune cell function change in non-tumor lesions, studies based on primary pulmonary hypertension and sarcoidosis have shown that PD1-positive CD4+ cells exhibit a process of promoting fibrosis. Therefore, blocking PD1 antibody can inhibit and improve pulmonary fibrosis. These data suggest that PD1 positive cells are involved in the pathologic process of pulmonary fibrosis. Preliminary data showed that PD1 expression levels were differentiated in peripheral blood of patients with acute myocardial infarction. Further study on the expression and corresponding role of PD1/PD-L1 signaling pathway in ventricular remodeling may provide a new target for the treatment of myocardial infarction remodeling.

This is a perspective, self-controlled cohort study. This study aims to Compare high PD1+ T cell and low PD1+ T cell expression in peripheral blood for cardiac function prognosis in Patients with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age;
2. Understand oral confirm to accept the risks and benefits of this experiment could bring He (she) or its legal representative in experiment related to provide written informed consent before surgery;
3. Was diagnosed with st-elevation acute myocardial infarction;
4. Based on the visual assessment of coronary angiography of coronary artery stenosis degree is 50% and the row stenting patients;
5. The target vessels are limited to the main coronary arteries (including the left anterior descending, left circumflex, and right coronary arteries).

Exclusion Criteria:

1. Pregnant or lactating women; Patients with previous malignant tumors or mental diseases; Recent major trauma/trauma, or surgical treatment; Drug, drug and alcohol abusers; Those who have been receiving antitumor drugs, immunosuppressants, hormones and antibiotics for a long time; People with blood-borne infectious diseases (including hepatitis B, c, syphilis, AIDS, etc.);
2. People with immune deficiency diseases or autoimmune diseases; Liver and kidney dysfunction; Aortic dissection, pulmonary embolism, acute myocarditis or severe valvular disease; One who is in the acute phase of any illness (influenza, pneumonia, gastroenteritis, skin disease, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the department of Cardiology with a diagnosis of ST-segment elevation acute myocardial infarction, angiography indicating 50% stenosis of at least one major coronary artery and stent implantation were selected
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac function(echocardiography) recovery after 1 and 3 months was measured compared with baseline(at admission). | at admission, 1 month , 3 months
  Compare the changes of ejection fraction（%） at 1 and 3 months with baseline(at admission)

SECONDARY OUTCOMES:
Patient-oriented composite outcome | 3 months
  Patient-oriented composite outcome (POCO), defined as a composite of all death, myocardial infarction (MI) or any revascularization at 3 months according to the ARC definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD, PhD, Study Chair — 2nd Affiliated Hospital, School of Medicine at Zhejiang University; Xinyang Hu, MD, PhD, Study Director — 2nd Affiliated Hospital, School of Medicine at Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided